CLINICAL TRIAL: NCT02830438
Title: Shear Wave Elastography in Native Kidney Disease: a Pilot Study
Brief Title: Shear Wave Elastography in Native Kidney Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough participants recruited
Sponsor: Albert Einstein Healthcare Network (Other)
Responsible Party: Principal Investigator, Mario Naranjo-Tovar, MD, Principal Investigator, Albert Einstein Healthcare Network
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 4837; 8574 (Other Grant/Funding Number: Albert Einstein Society Grant)
Record Dates: First submitted 2016-07-07; First posted 2016-07-12 (Estimated); Results first posted 2020-06-05 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-05

CONDITIONS: Acute Kidney Disease; Chronic Kidney Disease
Keywords: kidney disease; fibrosis; ultrasound; elastography
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Shear wave elastography group (Experimental): Patients referred for kidney biopsy will then undergo shear wave elastography measurements.
  Interventions: Device: Shear wave elastography

INTERVENTIONS:
Device: Shear wave elastography — Ultrasound technique of the kidneys to assess wave elastography.

SUMMARY:
In this proposal, the aim is to examine shear wave elastography (SWE) measurements in diseased native kidneys and correlate them with grades of fibrosis using histological samples.

The overall goals of the proposed study are addressed by the following specific aim.

Specific aim: To determine whether differences exist in elasticity measurements between native kidneys with and without fibrosis.

Hypothesis: Kidneys with higher grades of fibrosis will demonstrate higher measures of tissue elasticity and stiffness compared to kidneys with zero fibrosis.

DETAILED DESCRIPTION:
The proposed project is a prospective cross-sectional study correlating native kidney shear wave elastography (SWE) measurements with histology. Briefly, patients referred for a native kidney biopsy will undergo SWE and the shear wave velocity (SWV) will be correlated with degree of fibrosis determined by a pathologist.

A list of patients who recently underwent a native kidney biopsy will be obtained from the pathology department on a weekly basis. Patients will then be contacted about participating in the study and consented during a follow up visit with their nephrologist.

After their biopsies, patients will be scheduled to come for a renal ultrasound and SWE. SWE examination will be conducted using an ultrasound machine equipped with a Philips Epiq ARFI Shear wave ElastPQ C1-5 mHz transducer. Shear wave velocity will be obtained and an estimate of tissue elasticity (Young's modulus) will be calculated. All measurements will be performed by one of two qualified radiology physicians who will be blinded to the clinical and pathological data. We will allow a period of 90 days to obtain the images after the biopsy; otherwise the patient is no longer eligible to participate.

The primary outcome measure of this study is to determine whether tissue elasticity determined by SWE can assess kidney fibrosis. Linear regression analysis will be performed to describe the relation of the extent of fibrosis and parenchymal stiffness.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years of age who are referred for a native kidney biopsy.

Exclusion Criteria:

* BMI > 35
* Patients with polycystic kidney disease, renal cell carcinoma, hydronephrosis or renal stones.
* Patients who develop severe post biopsy complications (infection, significant bleeding requiring transfusion or intervention)
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-06-10 (Actual); Study Completion 2018-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario Naranjo-Tovar, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu Q, Wang XY, He HG, Wei HM, Kang LK, Qin GC. Acoustic radiation force impulse imaging for non-invasive assessment of renal histopathology in chronic kidney disease. PLoS One. 2014 Dec 29;9(12):e115051. doi: 10.1371/journal.pone.0115051. eCollection 2014. PMID 25546304
- [Result] Samir AE, Allegretti AS, Zhu Q, Dhyani M, Anvari A, Sullivan DA, Trottier CA, Dougherty S, Williams WW, Babitt JL, Wenger J, Thadhani RI, Lin HY. Shear wave elastography in chronic kidney disease: a pilot experience in native kidneys. BMC Nephrol. 2015 Jul 31;16:119. doi: 10.1186/s12882-015-0120-7. PMID 26227484
- [Result] Lee J, Oh YT, Joo DJ, Ma BG, Lee AL, Lee JG, Song SH, Kim SU, Jung DC, Chung YE, Kim YS. Acoustic Radiation Force Impulse Measurement in Renal Transplantation: A Prospective, Longitudinal Study With Protocol Biopsies. Medicine (Baltimore). 2015 Sep;94(39):e1590. doi: 10.1097/MD.0000000000001590. PMID 26426636

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Outpatient
Period: Overall Study
Arm/Group | Shear Wave Elastography Group
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Shear Wave Elastography Group
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 52.1 [33 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 3
  Caucasian | 2
  Hispanic/Latino | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Shear Wave Velocity of Kidney Parenchyma
Description: The shear wave velocity of the kidneys will be determined using the elastography ultrasound machine. This will enable us to calculate the tissue elasticity using a standard formula. Shear wave velocity is measured in meters per second, at a range of 0-5 m/s with the highest number reporting hard consistency (fibrosis - worse outcome).
Time Frame: 6 months
Measure: Median (Standard Deviation); unit: meters per second
Arm/Group | Shear Wave Elastography Group
Number analyzed (Participants) | 8
meters per second | 0.21 (0.71)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Shear Wave Elastography Group
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed due to technical problems during recruitment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-05-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT02830438/Prot_SAP_000.pdf